CLINICAL TRIAL: NCT01088841
Title: The Functional Significance of Gut-expressed Taste Receptors in the Secretion of Glucagon-like Peptide-1 and Peptide YY
Brief Title: Sweet Taste Receptors and the Secretion of Glucagon-like Peptide-1 and Peptide YY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Beglinger Christoph, Prof. Dr. med., Department of Gastroenterology, University Hospital Basel, Basel, Switzerland
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EKBB 69/04.01
Record Dates: First submitted 2010-03-16; First posted 2010-03-17 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2011-02

CONDITIONS: Appetite and General Nutritional Disorders; Hormone Replacement
MeSH Terms: interventions — lactisole; Glucose; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 75 g glucose + 150 ppm lactisole (Active Comparator)
  Interventions: Dietary Supplement: lactisole
- 75 g glucose + 300 ppm lactisole (Active Comparator)
  Interventions: Dietary Supplement: lactisole
- 75 g glucose + 450 ppm lactisole (Active Comparator)
  Interventions: Dietary Supplement: lactisole
- 75 g glucose (Placebo Comparator)
  Interventions: Dietary Supplement: lactisole

INTERVENTIONS:
Dietary Supplement: lactisole — lactisole (flavoring agent/sweet taste antagonist) dissolved with 75 g glucose in 300 mL tap water; administered via intragastric tube
  Other Names: Glucose; water

SUMMARY:
The purpose of this study is to determine the functional significance of sweet taste receptors in the secretion of GI satiety peptides by using a specific sweet taste receptor antagonist to block sweet taste perception in the gut.

DETAILED DESCRIPTION:
There is strong evidence that taste signaling mechanisms identified in the oral epithelium also operate in the gut. It is suggested that open-type enteroendocrine cells directly sense nutrient via alpha-gustducin coupled taste receptors to modulate the secretion of glucagon like peptide-1 (GLP-1) and peptide YY (PYY). Several nutrient responsive G-protein coupled receptors have been identified in the human gut, including the sweet taste responsive T1R2/T1R3 heterodimer, the amino acid/umami responsive T1R1/T1R3 as well as GPR120 for unsaturated long-chain free fatty acids.The functional significance of sweet taste receptors in glucose stimulated secretion of GLP-1 and PYY will be determined by intragastric infusion of 75 g glucose with different concentrations of lactisole (150 ppm, 300 ppm and 450 ppm)in a double blind, 4-way crossover trial including 16 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* BMI of 19.0-24.5
* Age 18-40
* stable body weight for at least 3 month

Exclusion Criteria:

* smoking
* substance abuse
* regular intake of medication
* medical or psychiatric illness
* gastrointestinal disorders or food allergies

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal peptide secretion | 2 hours blood sampling

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Principal Investigator — Clinical Research Center, University Hospital Basel
Locations (1):
- University Hospital Basel, Clinical Research Center, Basel, Switzerland